CLINICAL TRIAL: NCT00337649
Title: An Open-label Study to Evaluate the Effect of Combination Therapy With Epothilone D and Herceptin on Tumor Response in Patients With HER-2 Overexpressing Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Epothilone D in Combination With Herceptin (Trastuzumab) in Patients With HER-2 Positive Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NO17328
Record Dates: First submitted 2006-06-15; First posted 2006-06-16 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — desoxyepothilone B; Trastuzumab

ARMS (2):
- Phase I - Epothilone D Dose Escalation (Experimental)
  Interventions: Drug: Epothilone D; Drug: Herceptin
- Phase II - Epothilone D Maximum Tolerated Dose (Experimental)
  Interventions: Drug: Epothilone D; Drug: Herceptin

INTERVENTIONS:
Drug: Epothilone D — ≤100 mg/m^2 intravenously (iv) on days 1, 8 and 15 once every 4 weeks
  Other Names: RO4598715; KOS-862
Drug: Herceptin — 4mg/kg iv loading dose, followed by 2mg/kg iv weekly
  Other Names: Trastuzumab

SUMMARY:
This single arm study will determine the efficacy and safety of an epothilone D and Herceptin combination regimen in patients with HER-2 positive locally advanced or metastatic breast cancer. Epothilone D will be administered intravenously on days 1, 8 and 15 every 4 weeks at a dose not exceeding 100mg/m2. Herceptin will be administered intravenously on a weekly schedule; a 4mg/kg loading dose will be followed by a weekly maintenance dose of 2mg/kg. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* women >=18 years;
* locally advanced or metastatic breast cancer;
* HER-2 overexpression (FISH + or IHC 3+);
* >=1 measurable lesion;
* up to one prior anthracycline-based chemotherapy regimen in a metastatic setting.

Exclusion Criteria:

* pre-existing neuropathy >=grade 2;
* known CNS metastases;
* congestive heart failure, or myocardial infarction within the last 6 months;
* previous malignancies in last 5 years, except for cured basal cell cancer of the skin, or cancer in situ of the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2004-05; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Phase I: Number of Participants with a Dose-Limiting Toxicity | From first dose of study treatment until end of Cycle 1 (1 cycle is 28 days)
Phase II: Objective Response Rate (per RECIST criteria) | From first dose of study treatment until documented response (up to 3 years, 2 months)

SECONDARY OUTCOMES:
Phase II: Duration of Response | From date of objective response until progressive disease or death, whichever occurs first (up to 3 years, 2 months)
Phase II: Time to Tumor Progression | From first dose of study treatment until progressive disease or death, whichever occurs first (up to 3 years, 2 months)
Phase I: Plasma Concentration of Epothilone D at Specified Timepoints | Cycle 1 Days -2, -1, and 1; Cycle 2 Days 1 15-17 (1 cycle is 28 days)
Number of Participants with at Least One Adverse Event | From first dose of study treatment until 28 days after last dose (up to 3 years, 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- Spain (3):
  - Barcelona
  - Madrid
  - Valencia